CLINICAL TRIAL: NCT02749383
Title: A Randomized, Double-blind, Single Center, Investigator-initiated Clinical Study to Evaluate the Safety and Efficacy of PAC-14028 Cream in Subjects With Mild to Moderate Seborrheic Dermatitis of the Face
Brief Title: A Study to Evaluate the Safety and Efficacy of PAC-14028 Cream in Seborrheic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amorepacific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TRPV1-SD_IIT
Record Dates: First submitted 2015-09-30; First posted 2016-04-25 (Estimated); Last update posted 2016-04-25 (Estimated); Status verified 2016-04

CONDITIONS: Seborrheic Dermatitis
MeSH Terms: conditions — Dermatitis, Seborrheic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- PAC-14028 cream 0.3% (Experimental): Twice daily for 4 weeks
  Interventions: Drug: PAC-14028 cream 0.3%
- PAC-14028 cream 1.0% (Experimental): Twice daily for 4 weeks
  Interventions: Drug: PAC-14028 cream 1.0%
- PAC-14028 cream vehicle (Placebo Comparator): Twice daily for 4 weeks
  Interventions: Drug: PAC-14028 cream vehicle

INTERVENTIONS:
Drug: PAC-14028 cream 0.3% — Topical application
  Arms: PAC-14028 cream 0.3%
Drug: PAC-14028 cream 1.0% — Topical application
  Arms: PAC-14028 cream 1.0%
Drug: PAC-14028 cream vehicle — Topical application
  Arms: PAC-14028 cream vehicle

SUMMARY:
This study is a Phase II, single center, randomized, double-blind, placebo-controlled study in male and female subjects, aged ≥ 19 years with mild to moderate seborrheic dermatitis of the face. All subjects will receive BID topical applications of PAC-14028 cream or vehicle for up to 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged between 19 and 65 years old
* Clinical diagnosis of seborrheic dermatitis in the facial area with Erythema severity ≥ 2 and Scaling severity ≥ 2
* IGE (Investigator's Global Evaluation) Score 2 or 3

Exclusion Criteria:

* Patients with psoriasis, atopic dermatitis, facial acne, rosacea or perioral dermatitis
* Patients who have been infected with bacteria, fungi, virus and animal infectious disease on the facial area
* Patients who were administered topical antifungal agents, steroids, retinoids, or calcineurin suppressants for the treatment of seborrheic dermatitis within the last 2 weeks
* Patients who were administered systemic antifungal agents, steroids, retinoids, or immunosuppressants for the treatment of seborrheic dermatitis within the last 4 weeks
* Patients who were administered local antibiotics for the treatment of seborrheic dermatitis within the last 4 weeks
* Pregnant women, breastfeeding women or women of childbearing potential or women who are planning a pregnancy during the study

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2014-02; Primary Completion 2014-12 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Treatment success rate in IGE(Investigator's Global Evaluation) | Change from Baseline at Day 14 and Day 28
  Treatment success rate in IGE on 28th day from the baseline

SECONDARY OUTCOMES:
Change in Erythema severity score | Change from baseline at Day 14 and 28
Change in Scale severity score | Baseline, Day 14 and Day 28
  Change from baseline at Day 14 and 28
Change in Visual Analogue Scale(VAS) score | Change from baseline at Day 14 and 28

CONTACTS AND LOCATIONS:
Overall Officials: BeomJoon Kim, Professor, Principal Investigator — Department of Dermatology, Chungang University Hospital